CLINICAL TRIAL: NCT00962325
Title: Increasing Physical Activity Among Inactive Bariatric Surgery Patients
Brief Title: Increasing Physical Activity Among Inactive Bariatric Surgery Patients (Bari-Active)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dale Bond, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK83438; K01DK083438 (NIH); DK083438-01; NCT00820066 (obsolete NCT alias)
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Physical Activity; Weight Loss; Health-related Quality of Life
Keywords: Physical activity; Obesity; Bariatric surgery; Weight Loss
MeSH Terms: conditions — Motor Activity; Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activity behaviors counseling (Experimental)
  Interventions: Behavioral: Intervention to increase physical activity
- Standard care control (No Intervention): 6 weeks of standard preoperative care

INTERVENTIONS:
Behavioral: Intervention to increase physical activity — This will be a 6-week preoperative intervention to increase structured walking activity. This will be accomplished through weekly individual face-to-face sessions involving tailored instruction in use of standard behavior change strategies such as self-monitoring, goal-setting, stimulus control, etc.
  Arms: Activity behaviors counseling

SUMMARY:
For the growing number of severely obese individuals, there are currently few effective long-term weight control options with the exception of bariatric surgery. However, behavioral factors including low physical activity can undermine successful surgical outcomes. This study will compare the effects of a behavioral physical activity intervention with a standard care control condition on changes in physical activity among inactive adult bariatric surgery patients.

DETAILED DESCRIPTION:
The proportion of Americans who are severly obese or more than 100 pounds overweight is rapidly increasing. This presents a significant public health challenge as severely obese individuals have a higher rate of comorbidities and exact a greater toll on the health care system than less obese persons. For these individuals, bariatric surgery is currently the treatment of choice for producing substantial and long-term weight loss, although outcomes vary. Low physical activity is one behavioral factor that undermines surgical success. However, structured behavioral interventions to increase physical activity in bariatric surgery patients have not been conducted.

This study involves a randomized controlled trial that compares the effects of a behavioral intervention to increase physical activity with a standard care control group on changes in physical activity among adult bariatric surgery patients with low physical activity. Eighty bariatric surgery patients will be assigned to 6 weeks of either preoperative: (1) intervention to increase physical activity or (2) standard care control. Participants in the intervention group will receive individual, face-to-face sessions involving tailored instruction in use of standard behavior change strategies such as self-monitoring, goal setting and stimulus control. The PA intervention will focus on increasing home-based walking exercise. Physical activity will be objectively measured for 7 consecutive days via accelerometry at baseline/pre-intervention, post-intervention, and 3- and 6-months postoperative follow-up. At each time point, the groups will be compared on total moderate-to-vigorous physical activity (MVPA) minutes and MVPA minutes occurring in bouts of 10 minutes or longer. This study will test whether the behavioral physical activity intervention produces greater increases in pre- and post-operative physical activity than standard care. The long-term goal of this research is to improve bariatric surgery outcomes through innovative behavioral strategies to increase physical activity.

ELIGIBILITY:
Inclusion Criteria:

* BMI equal to or greater than 40 or greater than or equal to 35 (in presence of significant comorbidities)
* Have elected to undergo Roux-en-Y gastric bypass or laparoscopic adjustable gastric banding
* Able to engage in activities of daily living
* Currently inactive, defined as less than 150 weekly minutes of moderate-to-vigorous physical activity in bouts of 10 minutes or more
* Obtainment of written consent from surgeon to participate

Exclusion Criteria:

* Unable to engage in activities of daily living
* Report conditions that would render the participant unlikely to follow the study protocol (e.g., relocation, substance abuse, severe psychiatric condition)
* Inability to understand program instructions due to language barrier or a mental disability

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2014-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in MVPA minutes, bout-related (occurring in bouts of 10 minutes or longer) and total | 6-week Post-intervention follow-up

SECONDARY OUTCOMES:
Change in MVPA, bout-related and total | 3- and 6-month postoperative follow-up
Changes in health-related quality of life | 6-week Post-intervention follow-up, 3- and 6-month postoperative follow-up
Changes in physical activity self-efficacy and outcome expectations | Post-intervention follow-up, 3- and 6-month postoperative follow-up
Changes in physical activity enjoyment | Post-intervention, 3- and 6-month postoperative follow-up
Weight | post-intervention follow-up, 3- and 6-months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Dale s Bond, Ph.D., Principal Investigator — The Miriam Hospital/Brown Alpert Medical School
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Bond DS, Raynor HA, Thomas JG, Unick J, Webster J, Ryder B, Vithiananthan S. Greater Adherence to Recommended Morning Physical Activity is Associated With Greater Total Intervention-Related Physical Activity Changes in Bariatric Surgery Patients. J Phys Act Health. 2017 Jun;14(6):492-498. doi: 10.1123/jpah.2016-0529. Epub 2017 Mar 2. PMID 28253045
- [Derived] Bond DS, Vithiananthan S, Thomas JG, Trautvetter J, Unick JL, Jakicic JM, Pohl D, Ryder BA, Roye GD, Sax HC, Wing RR. Bari-Active: a randomized controlled trial of a preoperative intervention to increase physical activity in bariatric surgery patients. Surg Obes Relat Dis. 2015 Jan-Feb;11(1):169-77. doi: 10.1016/j.soard.2014.07.010. Epub 2014 Jul 30. PMID 25304832